CLINICAL TRIAL: NCT05284201
Title: Safety and Performance Assessment of the LIFT System When Used to Support Home-based Upper Extremity Training in Individuals With Spinal Cord Injury.
Brief Title: LIFT Home Study of Non-Invasive ARC Therapy for Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ONWARD Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DOC2530; Pro00059716 (Other: Advarra)
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Chronic Spinal Cord Injury
Keywords: SCI, Tetraplegia, ARC therapy
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Functional task practice and ARC Therapy (Experimental): FTP and ARC Therapy with the LIFT System at home for 1 month.
  Interventions: Device: LIFT System

INTERVENTIONS:
Device: LIFT System — The LIFT System delivers the Functional task practice and ARC Therapy to improve upper extremity function in individuals with tetraplegia.

SUMMARY:
The LIFT Home Study is an observational, single-arm study designed to assess the safety of non-invasive electrical spinal stimulation (ARC Therapy) administered by the LIFT System to treat upper extremity functional deficits in people with chronic tetraplegia.

DETAILED DESCRIPTION:
The primary goal of this study is to report on the safety of the study device when used at home. In addition, the study will report on observed changes in upper extremity function and strength after a period of home use.

The LIFT Home Study will enroll subjects who have recently completed participation in the Up-LIFT Study. The study includes a set of baseline assessments to be completed in the clinic, a four-week home use treatment program prescribed by the investigator, and a final set of clinic-based assessments at the end of the study.

At the baseline visit, the subject and caregiver will be trained on the use of the device and prescribed a specific training regime for its use at home. The subject will be issued a device that is uniquely programmed to operate within a limited set of parameters as specified by the investigator.

Throughout the study, subjects will be prompted to report all adverse events (AE) regardless of relatedness to the device.

At baseline and the final clinic visit, UE strength and function will be measured with stimulation off using a comprehensive set of assessment tools including CUE-T, GRASSP, Pinch and Grasp Force, as well as patient and caregiver global impression of change questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. At least 22 years old and no older than 75 years old at the time of enrollment
2. Non-progressive cervical spinal cord injury from C2-C8 inclusive
3. American Spinal Injury Association (ASIA) Impairment Scale (AIS) classification B, C, or D
4. Indicated for upper extremity training procedures by subject's treating physician, occupational therapist or physical therapist
5. Minimum 12 months post-injury
6. Capable of providing informed consent
7. Completed the Up-LIFT Study within the prior 12 months

Exclusion Criteria:

1. Has uncontrolled cardiopulmonary disease or cardiac symptoms as determined by the Investigator
2. Has any unstable or significant medical condition that is likely to interfere with study procedures or likely to confound study endpoint evaluations like severe neuropathic pain, depression, mood disorders or other cognitive disorders
3. Has been diagnosed with autonomic dysreflexia that is severe, unstable, and uncontrolled
4. Requires ventilator support
5. Has an autoimmune etiology of spinal cord dysfunction/injury
6. Spasms that limit the ability of the subjects to participate in the study training as determined by the Investigator
7. Breakdown in skin area that will come into contact with electrodes
8. Has any active implanted medical device
9. Pregnant, planning to become pregnant or currently breastfeeding
10. Concurrent participation in another drug or device trial that may interfere with this study
11. In the opinion of the investigators, the study is not safe or appropriate for the participant

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Incidence of all adverse events (AEs) | Through completion of the study, an average of 6 months
  Observational data regarding the incidence of all adverse events related to the use of the study device and treatment procedures will be reported.

SECONDARY OUTCOMES:
Extended use of the LIFT System at home | Through completion of the study, an average of 6 months
  The secondary outcome measure will report on the potential for extended use of the LIFT System at home to sustain or advance performance gains achieved during the prior in-clinic treatment phase. Upper extremity performance will be assessed using the CUE-T, GRASSP, Pinch and Grasp Force assessments and the Global Impression of Change questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Candace Tefertiller, PT, DPT, PhD, NCS, Principal Investigator — Craig Hospital, Colorado, United States
Locations (5):
- United States (5):
  - Craig Hospital, Englewood, Colorado
  - Shepherd Center- Crawford Research Institute, Atlanta, Georgia
  - INSPIRE Laboratory, Spaulding Hospital, Cambridge, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inanici F, Samejima S, Gad P, Edgerton VR, Hofstetter CP, Moritz CT. Transcutaneous Electrical Spinal Stimulation Promotes Long-Term Recovery of Upper Extremity Function in Chronic Tetraplegia. IEEE Trans Neural Syst Rehabil Eng. 2018 Jun;26(6):1272-1278. doi: 10.1109/TNSRE.2018.2834339. PMID 29877852
- [Background] Hoffman L, Field-Fote E. Effects of practice combined with somatosensory or motor stimulation on hand function in persons with spinal cord injury. Top Spinal Cord Inj Rehabil. 2013 Fall;19(4):288-99. doi: 10.1310/sci1904-288. PMID 24244094
- [Derived] Tefertiller C, Trumbower RD, Morse L, Pradarelli J, Gelenitis K, D'Amico JM, Moritz C, Field-Fote EC. Home-Based Noninvasive Spinal Cord Stimulation Safely Enhances Hand and Arm Function in People With Spinal Cord Injury. Neurol Clin Pract. 2025 Dec;15(6):e200537. doi: 10.1212/CPJ.0000000000200537. Epub 2025 Sep 24. PMID 41019097